CLINICAL TRIAL: NCT00380003
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Crossover Study to Assess the Efficacy of Two Doses of EVT 201 in the Treatment of Primary Insomnia in Adult Patients
Brief Title: Efficacy Study of EVT 201 to Treat Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evotec Neurosciences GmbH (Industry)
Organization: Evotec International GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — EVT 201

INTERVENTIONS:
Drug: EVT 201

SUMMARY:
The purpose of this study is to determine whether a compound known as EVT 201 is effective in treating people diagnosed with primary insomnia ( difficulty sleeping with no other significant contributing factor, such as depression).

ELIGIBILITY:
Inclusion Criteria:

* must have a diagnosis of primary insomnia
* over the last three months, must have a normal bedtime of between 9 pm and 1 am and a time in bed of at least 7 hours
* must be able to attend the Sleep Center for two consecutive nights on four occasions over a two month period
* must be willing and able to complete a sleep diary and questionnaires

Exclusion Criteria:

* must not have a clinically significant or unstable medical condition that may interfere with sleep
* must not have a major psychiatric disorder (other than insomnia) such as depression, schizophrenia, bipolar disorder
* must not be currently using any medication know to affect sleep e.g. hypnotics, anxiolytics,antidepressants, antihistamines, anticonvulsants
* must not intentionally nap 3 (or more) times per week
* must not smoke more than 10 cigarettes per day and /or be able not to smoke without distress or discomfort for the duration of visits to the sleep laboratory ( i.e. approximately 12 hours)

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time
Wake after sleep onset

SECONDARY OUTCOMES:
Latency to persistent sleep
Number of awakenings
Total wake time
Minutes of stages 1-4 and REM sleep
REM latency
Patient reported sleep variables
Residual sedation measures
Safety assessments including adverse events, ECgs, vital signs and routine laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: James K Walsh, PhD, Principal Investigator — St. Luke's Hospital, Sleep Medicine and Research Center, Chesterfield, MI
Locations (5):
- United States (5):
  - St Petersburg Sleep Disorders Center, St. Petersburg, Florida
  - The Sleep Disorders Center of Georgia, Peachtree Dunwoody Medical Center,5505 Peachtree Dunwoody Road, Suite 548, Atlanta, Georgia
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - St. Luke's Hospital, Chesterfield (St Louis), Missouri
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio